CLINICAL TRIAL: NCT02899039
Title: Follicular Helper T Cells: Biological Marker and Involvement in the Physiopathology of the IgG4-related Disease
Acronym: G4-FH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-31; RC12_3608 (Registry Identifier: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2016-09

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IgG4-related disease (Experimental): Subjects suffering from IgG4-related disease
  Interventions: Biological: extra blood draw samples
- Sjögren syndrome (Active Comparator): Subjects suffering from Sjôgren syndrome
  Interventions: Biological: extra blood draw samples
- Healthy controls (Active Comparator): Healthy subjects
  Interventions: Biological: extra blood draw samples

INTERVENTIONS:
Biological: extra blood draw samples

SUMMARY:
IgG4-related disease is a rare and very recently identified pathology, whose frequency is certainly underestimated.

The clinical presentation varies among affected organs, and most often, patients have at least three organ damage.

These organs exhibit tissue infiltration mononuclear polymorphic cells with often severe fibrosis progression resulting in a loss of function.

The biomarker, though not specific, is a polyclonal elevated serum IgG4, and histological marker, currently held by several teams, is the presence within the inflammatory infiltrate, of a predominance of IgG4-expressing plasma-cells with a relative plasma-cells IgG4 + / IgG +> 50% on tissue immunostaining.

The investigators project provides a global assessment of T lymphocyte abnormalities and specifically the TFH (Follicular Helper) during this IgG4-related disease compared to so-called groups "control" subjects suffering from Sjogren syndrome or healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* IgG4-related disease patients or
* Sjogren syndrome patients or
* Healthy subjects

Exclusion Criteria:

* Presence of autoimmune or inflammatory associated disease
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-07-17; Primary Completion 2015-05-04 (Actual); Study Completion 2016-05-07 (Actual)

PRIMARY OUTCOMES:
Proportion of Follicular Helper T cells (CD4 + CXCR5 + ICOShigh) in the blood | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- APHM, Marseille, France